CLINICAL TRIAL: NCT03623113
Title: The Dietary Education Trial in Carbohydrate Counting (DIET-CARB Study): A Randomized, Parallel, Open-label, Intervention Study Comparing Different Approaches to Dietary Self-management in Patients With Type 1 Diabetes
Brief Title: The Dietary Education Trial in Carbohydrate Counting (DIET-CARB Study in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bettina Ewers, Head of Nutrition, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18014897
Record Dates: First submitted 2018-07-19; First posted 2018-08-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Type1diabetes; Type1 Diabetes Mellitus; Glucose Metabolism Disorders
Keywords: Carbohydrate counting; Basic carbohydrate counting; Advanced carbohydrate counting; Carbohydrates; Diet
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCC intervention (Experimental): The BCC program consists of three group sessions and is delivered by two trained dietitians. In addition to the BCC program, the participants receive regular medical care in the diabetes clinic
  Interventions: Behavioral: BCC intervention
- ABC-ACC intervention (Experimental): The ABC-ACC program consists of one group session and two individual follow-up sessions and is delivered by trained dietitians with supervision by a medical doctor. In addition to the ABC-ACC program, the participants receive regular medical care in the diabetes clinic
  Interventions: Behavioral: ABC-ACC intervention
- Standard dietary education (Active Comparator): The routine outpatient dietary care consists of three individual consultations delivered by a trained dietitian. The individual guidance is based on the overall treatment goal(s), the defined personal dietary goals for behavioral change which will be in accordance with the patient's needs and preferences. In addition to the dietary counselling, the participants receive regular medical care in the diabetes clinic
  Interventions: Behavioral: Standard dietary education

INTERVENTIONS:
Behavioral: BCC intervention — Structured training and education i basic carbohydrate counting principles
  Other Names: Basic carbohydrate counting
  Arms: BCC intervention
Behavioral: ABC-ACC intervention — Structured training and education i advanced carbohydrate counting principles including the use of a automated bolus calculator carbohydrate
  Other Names: Advanced carbohydrate counting with a bolus calculator
  Arms: ABC-ACC intervention
Behavioral: Standard dietary education — Personalized individual dietary counselling based on overall meal planning, dietary guidelines and the patient's need and preferences
  Other Names: Routine dietary care
  Arms: Standard dietary education

SUMMARY:
The study is designed to evaluate two different dietitian-led self-management approaches in carbohydrate counting compared to routine dietary care (control) on glycaemic control in adult patients with type 1 diabetes:

1. The basic carbohydrate counting concept aims at improving carbohydrate counting accuracy and day-to-day consistency of carbohydrate intake (the BCC intervention)
2. The advanced carbohydrate counting concept aims at improving prandial insulin dose accuracy using an automated bolus calculator (the ABC-ACC intervention)

The main hypothesis is that structured training and education in either the BCC concept or the ABC-ACC concept will reduce HbA1c or the average glucose variability more than routine dietary education.

DETAILED DESCRIPTION:
The current study is a randomized controlled trial with a parallel-group design. A total of 231 patients will be enrolled in the trial. Participants will be randomized to one of three arms: 1) Basic carbohydrate counting (BCC), 2) Advanced carbohydrate counting with an automated bolus calculator (ABC-ACC), or 3) Standard dietary care.

The primary objective is to evaluate the six months effects of education in the BCC concept and the ABC-ACC concept compared to standard dietary care on glycaemic control as assessed by HbA1c or MAGE (mean amplitude of glycaemic excursions).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Diabetes duration; >12 months
* HbA1c of 53-97 mmol/mol
* Multiple daily insulin injection therapy
* Provided voluntary written informed consent

Exclusion Criteria:

* Practicing carbohydrate counting, as judged by the investigator
* Participated in a BCC group program within the last two years
* Use of insulin pump, or plans of having an insulin pump within the study period
* Fixed dose of rapid acting insulin therapy for meals
* Split-mixed insulin therapy
* Use of open CGM
* Use of Freestyle Libre
* Use of an automated bolus calculator
* Gastroparesis
* Pregnancy or breastfeeding, or plans of pregnancy within the study period
* Low daily intake of carbohydrates (defined as below 25 E% or 100 g/day), as judged by the investigator
* Uncontrolled medical issues, as judged by the investigator or a medical expert
* Concomitant participation in other clinical studies
* Unable to understand the informed consent and the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 6 months
  mmol/mol
Change in mean amplitude of glycaemic excursions (MAGE) | Baseline, 6 months
  mmol/l

SECONDARY OUTCOMES:
Change in HbA1c | 12 months
  mmol/mol
Change in body weight | Baseline, 6 months, 12 months
  kg
Change in low-density lipoprotein cholesterol (LDL-C) | Baseline, 6 months, 12 months
  mmol/l
Change in high-density cholesterol (HDL-C) | Baseline, 6 months, 12 months
  mmol/l
Change in total cholesterol (TC) | Baseline, 6 months, 12 months
  mmol/l
Change in free fatty acids (FFA) | Baseline, 6 months, 12 months
  mmol/l
Change in triglycerides (TG) | Baseline, 6 months, 12 months
  mmol/l
Change in systolic blood pressure | Baseline, 6 months, 12 months
  mm Hg
Change in diastolic blood pressure | Baseline, 6 months, 12 months
  mm Hg
Change in waist circumference | Baseline, 6 months, 12 months
  cm
Change in hip circumference | Baseline, 6 months, 12 months
  cm
Change in total fat free mass | Baseline, 6 months
  gram
Change in total fat mass | Baseline, 6 months
  gram
Change in time in range (3.9-10.0 mmol/l) | Baseline, 6 months
  Percent (%)
Changes in % time spent in hypoglycaemia (<3.9 mmol/l) | Baseline, 6 months
  Percent (%)
Change % time spent in hyperglycaemia (e.g. >11.1 mmol/l) | Baseline, 6 months
  Percent (%)
Change in standard deviation of mean plasma glucose | Baseline, 6 months
  mmol/l
Change in mathematical literacy | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in carbohydrate estimation accuracy | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in diet-related quality of life | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in perceived competences in diabetes | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in degree of autonomy-supportive dietitian | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in total energy intake | Baseline, 6 months
  kJ/day
Change in dietary intake of carbohydrates | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of total fat | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of saturated fatty acids (SFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of monounsaturated fatty acids (MUFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of polyunsaturated fatty acids (PUFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of protein | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of added sugar | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in intake of dietary fibre | Baseline, 6 months
  gram/day or g/MJ

OTHER OUTCOMES:
Change in physical activity level | Baseline, 6 months, 12 months
  Total score or percent (%)
Change in urinary biomarkers of carbohydrate intake | Baseline, 6 months
  Percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Ewers, MSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ewers B, Vilsboll T, Andersen HU, Bruun JM. The dietary education trial in carbohydrate counting (DIET-CARB Study): study protocol for a randomised, parallel, open-label, intervention study comparing different approaches to dietary self-management in patients with type 1 diabetes. BMJ Open. 2019 Sep 3;9(9):e029859. doi: 10.1136/bmjopen-2019-029859. PMID 31481560

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03623113/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03623113/SAP_001.pdf